CLINICAL TRIAL: NCT04504591
Title: Validation Of A New S-ICD Algorithm To Reduce Oversensing Of Dynamic T-Waves In Patients With Brugada Syndrome
Acronym: DE-08-16
Status: Terminated | Type: Observational
Why Stopped: Early termination due to COVID19; preliminary data can be considered significant
Sponsor: Angelo Auricchio (Other)
Responsible Party: Sponsor-Investigator, Angelo Auricchio, Prof., Cardiocentro Ticino
Organization: Cardiocentro Ticino (Other)
Other Study IDs: DE-08-16
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Brugada Syndrome 1S

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study will be to assess the efficacy of S-ICD with SMART Pass to discriminate dynamic T-waves amplitudes and morphologies over time.

Pilot, multi-centric, prospective, blinded, one arm (repeated measures), non-interventional study. Objective is to setup a 8-center data collection registry between Switzerland, Italy and Belgium.

DETAILED DESCRIPTION:
The subcutaneous implantable cardioverter-defibrillator (S-ICD) should be considered as an alternative to transvenous defibrillators in patients with an ICD indication when pacing therapy for bradycardia support, cardiac resynchronization or ventricular tachycardia management is not necessary.1 This class IIa recommendation from the 2015 ESC guidelines can often be applied to patients with inherited channelopathies, since these patients usually require decades of ICD therapy without developing a need for any type of pacing support. On the other hand, especially in patients with Brugada Syndrome (BrS), the dynamic nature of ECG morphology may increase the risk for cardiac T-wave oversensing (TWOS), which has also been reported the main cause of inappropriate shocks (IAS) in the general S-ICD population. In order to avoid unnecessary sensing issues with the S-ICD, baseline ECG screening is recommended prior to the implantation procedure. Recently, it has been shown that eligibility failure for S-ICD can occur in up to 13% of patients with an inherited primary arrhythmia syndrome and that patients with BrS present the highest rate of screening failure if compared with other channelopathies.

As of yet, this QRS and T-wave morphology assessment can be done with an algorithm-based automated screening tool (AST) that mimics the sensing set-up process of the S-ICD after implant.

Recently, a novel 9Hz high-pass filter (SMART Pass, available for all EMBLEM S-ICD models) has been introduced to reduce the risk of TWOS with the S-ICD12. This algorithm is only available with the S-ICD sensing mechanism and has not been incorporated in the automated screening software12. Retrospective modelling of inappropriate shock events recorded in the EFFORTLESS registry have shown a reduction in inappropriate shocks by ~80% with SMART Pass compared to the first generation sensing algorithm of the S-ICD13. This was achieved without affecting the detection and the time to therapy for true ventricular arrhythmias.

Prospective data are lacking about the effectiveness of SMART Pass to discriminate T-waves in patients with dynamic ECG morphologies. This may be of particular interest since the occurrence of ECG morphology disturbances is usually difficult to be predicted in individual patients. As such, these data will provide additional guidance to the mandatory screening process for all S-ICD candidates, in particular for those who have a known risk factor for dynamic ECG changes, like patients withBrS. The main objective of this study will be to assess the efficacy of S-ICD with SMART Pass to discriminate dynamic T-waves amplitudes and morphologies over time.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects beyond the ages of ≥18 the time of informed consent;
2. Subjects with suspected BrS;

Exclusion Criteria:

1. Presence of baseline Brugada type I ECG
2. Presence of structural cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Consecutive patients with suspected BrS will be submitted for routine diagnostic ajmaline testing
Study Population: Consecutive patients with suspected BrS will be submitted for routine diagnostic ajmaline testing.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of S-ICD screening failure due to TWOS with and without SMART Pass in patients with ajmaline-induced Brugada Type I ECG. | through study completion, an average of 15 months
  Rate of S-ICD screening failure due to TWOS after ajmaline challenge with and without SMART Pass in patients with Ajmaline induced Brugada type I ECG.

SECONDARY OUTCOMES:
Rate of S-ICD screening failure with and without SMART Pass in the patients without ajmaline-induced Brugada type-I ECG who manifest a conduction disturbance (i.e. RBBB). | through study completion, an average of 15 months
  Rate of S-ICD screening failure due to TWOS after ajmaline challenge with and without SMART Pass in patients without Brugada type I EC but with Ajmaline induced ECG conduction disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Conte, Dr., Principal Investigator — Fondazione Cardiocentro Ticino
Locations (6):
- UZ-VUB Brussels, Brussels, Belgium
- Italy (3):
  - Azienda Ospedaliera Brotzu, Cagliari
  - ATS Sardegna Ospedale San Francesco-ASSL 3 NUORO, Nuoro
  - Fondazione I.R.C.C.S. Policlinico San Matteo di Pavia, Pavia
- Switzerland (2):
  - Hopitaux Universitaires de Genève, Geneva
  - Fondazione Cardiocentro Ticino, Lugano

REFERENCES:
- [Derived] Conte G, Cattaneo F, de Asmundis C, Berne P, Vicentini A, Namdar M, Scalone A, Klersy C, Caputo ML, Demarchi A, Ozkartal T, Salghetti F, Casu G, Passarelli I, Mameli S, Shah D, Burri H, De Ferrari G, Brugada P, Auricchio A. Impact of SMART Pass filter in patients with ajmaline-induced Brugada syndrome and subcutaneous implantable cardioverter-defibrillator eligibility failure: results from a prospective multicentre study. Europace. 2022 May 3;24(5):845-854. doi: 10.1093/europace/euab230. PMID 34499723